CLINICAL TRIAL: NCT04215419
Title: The Furosemide Stress Test, Electrolytes Response and Renal Index in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Hospital San Paolo (Other)
Responsible Party: Principal Investigator, Davide Chiumello, Professor, Hospital San Paolo
Other Study IDs: 2019/ST/094
Record Dates: First submitted 2019-12-20; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Acute Kidney Injury
Keywords: Kidney; Furosemide; Renal Index; Stress Test; sodium; Potassium; Chloride
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Urine sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of the present study is to compare the response to furosemide stress test in term of diuresis and electrolytes and of the renal index in mechanically ventilated patients at admission and after 3 days in patients with and without the presence of AKI

DETAILED DESCRIPTION:
The acute kidney injury (AKI) is a common clinical syndrome in critically ill patients, occurring in up of 60% of the patients, and almost 40% of these patients will die within 90 days . Between 5% to 10% of the patients with AKI requires renal replacement therapy and only 30% will be alive after 5 years . The most common reported contributing factors to AKI were sepsis, major surgery, cardiogenic shock, hypovolemia and potentially related drugs . Although the AKI has been classically defined as an abrupt and sustained decrease in renal function and is commonly assessed on serum creatinine rise and/or fall in urine output there are not clear cutoffs for the diagnosis . Unfortunately the changes in these two parameters are poor predicting of AKI in critically ill patients . In the recent years several renal biomarkers have been proposed to accurately detect acute tubular injury before serum creatinine changes with possible improvement in the outcome; however the evidence was quite low . Because the majority of early AKI are related to an acute tubular injury, it has been suggested to evaluate the tubular function reserve by a bolus of furosemide (i.e. the furosemide stress test). As an organic acid, furosemide is tightly bound to serum proteins and gains access to the tubular urinary space through active secretion in the proximal convoluted tubule via the human organic anion transporter system .Once in the tubular lumen, furosemide inhibits chloride transport throughout the thick ascending limb of Henle, preventing sodium reabsorption: this results in natriuresis, increased urine flow and potentially reduced tubular oxygen demand . Specially a relatively intact kidney, with preserved estimated glomerular filtration rate (eGFR) and tubular function, should respond to furosemide with a quick diuresis, whereas tubular injury can be associated with urine output that is relatively preserved at baseline, but that fails to significantly augment with a diuretic challenge. In one mixed (retrospective and prospective) study and in one randomized trial in critically ill patients admitted in intensive care with mild AKI, the furosemide stress test was able to predict the progression to severe AKI. Furthermore also the response to electrolyte excretion should predict the possible presence of AKI . In addition the renal imaging techniques by ultrasound, which are non invasive and repeatable, are considered a mandatory component of the AKI diagnostic work up . Among the available imaging technique the renal resistive index (RI) which compute the ratio between the systolic and diastolic blood velocity in the arcuate or interlobular arteries is the most common used due to the easiness and to the good reproducibility . Although the physiological and clinical significance of RI is still debated because is related to the resistance and compliance of the renal vessels and to the central hemodynamic , previous studies have shown the utility of RI to predict both the occurrence and the reversibility of AKI .

Aim of the present study is to compare the response to furosemide stress test in term in diuresis and electrolytes and of the renal index in mechanically ventilated patients at admission and after 3 days in patients with and without the presence of AKI

All consecutive mechanically ventilated patients, following an hemodynamic stabilization (mean arterial pressure of at least 65 mmHg without the need for fluid bolus and/or start or increase in the dose of vasopressors or inotropic drugs within the last 6 h), admitted to the General Intensive Care of Santi Paolo-Carlo Hospital were enrolled. Exclusion criteria were: an age < 18 years, pregnancy, hemodynamic instability (defined as mean arterial pressure (MAP)<60 mmHg), a suspected or confirmed obstructive renal failure, the presence of a chronic renal failure, as defined by a basal creatinine clearance value < 30 ml min-1 . During the study the level of sedation and the ventilatory setting were not changed.

Renal index

The renal index examination was performed by one among three dedicated physicians, who were not in charge of the patients and trained with ultrasound examinations . Doppler ultrasonography will be performed at the patient's bedside by the same trained operator using an ultrasound scanner (LogiQ7 General Electric Healthcare, UK) with a 5 Mega-hertz transducer. The Doppler measurements will be obtained from the right kidney in all patient. After visualization of the kidney in gray scale and color Doppler modes, the absence of signs of chronic renal damage will be checked. The interlobar or arcuate arteries will be localized with sonography and color Doppler mode. Blood velocities in the interlobar arteries will be recorded using pulse-wave Doppler. RI will be calculated as follow:

RI= (Peak Systolic velocity - end Diastolic Velocity)/Peak systolic velocity and average.

At least three readings will be obtained from the selected arteries, and the mean of the corresponding three renal RI determinations will be used for the study

Furosemide stress test After the ultrasonography evaluation, the patients will be tested with the Furosemide Stress Test (FST). Who will be loop-diuretic naïve will be given 1.0 mg/kg of intravenous furosemide. Because patients who are previously treated with loop diuretics within the previous 7 days are likely to have a blunted response over time compared to naïve patients, this group will receive an intravenous dose of 1.5 mg/kg) . In order to minimize the risk of hypovolemia, urine output will be replaced ml for ml each hour with Ringers lactate for six hours after the FST.

Data collection Before and after two hours of the renal index and the furosemide stress text the following clinical and laboratory data were collected: mean arterial pressure, central venous pressure, heart rate, plasma and urine amount of sodium, potassium, chloride, and arterial blood gas analysis. The urine volume was measured after one and two hours

ELIGIBILITY:
Inclusion Criteria:

* all mechanically ventilated patients

Exclusion Criteria:

* age < 18 years
* pregnancy
* hemodynamic instability (defined as mean arterial pressure (MAP)<60 mmHg)
* suspected or confirmed obstructive renal failure,
* presence of a chronic renal failure, as defined by a basal creatinine clearance value < 30 ml min-1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive mechanically ventilated patients, following an hemodynamic stabilization (mean arterial pressure of at least 65 mmHg without the need for fluid bolus and/or start or increase in the dose of vasopressors or inotropic drugs within the last 6 h), admitted to the General Intensive Care of Santi PaoloCarlo Hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2019-10-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Response to furosemide stress test in patients with and without AKI | Two hours after furosemide stress test
  Urine volume after furosemide administration,
Urine output of sodium, potassium and chloride after furosemide stress test | Two hours after furosemide stress test
  Determination of Urinary Sodium concentration (meq/L)

SECONDARY OUTCOMES:
Renal Index in patients with and without AKI | At admission
  Determination of the ratio between the systolic and diastolic blood velocity in the arcuate or interlobular kidney arteries

CONTACTS AND LOCATIONS:
Overall Officials: Davide Chiumello, Professor, Principal Investigator — ASST Santi Paolo e Carlo, ospedale San Paolo
Locations (1):
- ASST Santi Paolo Carlo Ospedale San Paolo, Milan, Italy

IPD SHARING:
Plan to Share IPD: No